CLINICAL TRIAL: NCT07398872
Title: Evaluating the Safety and Efficacy of AAV9.hMCOLN1co in Treating Mucolipidosis Type IV: A Single-Center, Interventional, Open-Label, Single-Arm Clinical Study
Brief Title: Safety and Efficacy of AAV9. hMCOLN1co For Patients With Mucolipidosis Type IV
Acronym: AAV9-hMCOLN1
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAV9. hMCOLN1co.01
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Mucolipidosis Type IV
Keywords: Mucolipidosis Type IV,; MLIV
MeSH Terms: conditions — Mucolipidoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm AAV9. hMCOLN1co, a gene therapy product (Experimental)
  Interventions: Biological: AAV9.hMCOLN1co

INTERVENTIONS:
Biological: AAV9.hMCOLN1co — A single intrathecal infusion of 10 mL at 2E13 vg/mL for a total dose of 2E14 vg

SUMMARY:
Safety and Efficacy of AAV9.hMCOLN1co for patients with Mucolipidosis Type IV(MLIV): A Single-Center, Interventional, Open-Label, Single-Arm Clinical Study. The goal of this clinical trial is to evaluate whether a gene therapy can safely treat children with MLIV.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between 1.5 and 8 years of age(inclusive) at the time of signing the informed consent form
2. Diagnosed with Mucolipidosis type IV caused by MCOLN1 gene mutations
3. The legal guardian and/or the participant(if applicable) has signed the informed consent form
4. Meet the criteria for anesthesia and sedation appropriate for their age(as assessed by the investigator)
5. Has completed age-appropriate immunizations according to the National Immunization Program Schedule for Children

Exclusion Criteria:

1. Presence of any contraindication to lumbar puncture or intrathecal therapy (e.g., spina bifida, meningitis, coagulation disorders, obstructive spinal internal fixation devices) or presence of a cerebrospinal fluid (CSF) diversion/shunting device
2. At screening, severe joint contracture as assessed by the physiotherapist, affecting functional assessment or intrathecal administration
3. X-ray examination indicating severe scoliosis (Cobb angle ≥ 50°)
4. History of, or planned, scoliosis corrective surgery within 1 year before or after dosing
5. Use of invasive respiratory support (e.g., tracheostomy with positive pressure ventilation) or oxygen saturation while awake < 95% (or < 92% at altitudes > 1000 m)
6. Requirement for ≥ 12 hours/day of non-invasive respiratory support within 2 weeks prior to dosing
7. Dependence on gastric tube feeding with the majority of nutrition taken non-orally, or body weight below the 3rd percentile for age according to World Health Organization (WHO) standards (patients with an existing gastrostomy are not excluded)
8. Active viral infection, including human immunodeficiency virus (HIV), hepatitis B, hepatitis C, etc.
9. In the investigator's judgment, occurrence of a serious non-respiratory infection (e.g., pyelonephritis, meningitis) within 4 weeks prior to dosing, or presence of other serious comorbid disease
10. In the investigator's judgment, severe renal and/or hepatic impairment
11. Known history of epilepsy, diabetes, idiopathic hypocalciuria, symptomatic cardiomyopathy, etc.
12. In the investigator's judgment, history of bacterial meningitis or central nervous system disease (including tumors), with MRI/computed tomography (CT) indicating abnormalities that may affect lumbar puncture or cerebrospinal fluid circulation
13. In the investigator's judgment, allergy to prednisolone or other glucocorticoids and their excipients
14. In the investigator's judgment, allergy to gadolinium or gadolinium-containing contrast agents
15. Concomitant use of medications for myopathy/neuropathy, antidiabetic drugs, immunosuppressants, plasma exchange, or immunomodulators (e.g., adalimumab), or receipt of immunosuppressive therapy (e.g., glucocorticoids, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, intravenous immunoglobulin, rituximab, etc.) within 3 months prior to dosing
16. Inability to discontinue laxatives or diuretics within 24 hours prior to dosing
17. Oral administration of β-receptor agonists within 30 days prior to dosing
18. Anti-AAV9 antibody titer > 1:50 (patients may be enrolled if a repeat test after a 2-4-week interval is ≤ 1:50)
19. Clinically significant abnormalities in laboratory parameters prior to gene replacement therapy, such as gamma-glutamyl transpeptidase (GGT)/ALT/AST/total bilirubin (TBIL) > 2 × upper limit of normal (ULN), estimated glomerular filtration rate (eGFR) < 60 mL/min, hemoglobin < 8 or > 18 g/dL, white blood cell count > 20,000/cmm, etc.
20. Anticipated need for major surgery (e.g., spinal surgery, tracheostomy) during the study period
21. Inability to comply with the study protocol or to attend scheduled follow-up visits
22. Refusal to sign the informed consent form and/or unwillingness to maintain the confidentiality of the study data.

Ages: 18 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2027-01-20 (Estimated); Study Completion 2031-01-20 (Estimated)

PRIMARY OUTCOMES:
To assess the types, severity, and incidence of adverse events(AEs) and serious adverse events(SAEs) following treatment | through study completion, an average of 5 years
  collection of occurrence and severity of serious adverse events. Incidence of serious adverse events and adverse events throughout the study, as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Higher grade values indicated greater severity. Grade 1 - Grade 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China